CLINICAL TRIAL: NCT05161286
Title: The Influence of Expectations, Attention and Test Paradigm on the Efficacy of the Pain Processing System
Brief Title: The Influence of Expectations, Attention and the Test Paradigm on the Efficacy of the Pain Processing System
Acronym: CPM_AWARE
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08516
Record Dates: First submitted 2021-08-12; First posted 2021-12-17 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-02

CONDITIONS: Pain
Keywords: endogenous pain modulation; conditioned pain modulation; expectations; attention; test paradigm
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy pain-free cohort: Healthy pain-free Dutch-speaking men and women between the age of 18 and 65 years

SUMMARY:
Conditioned pain modulation (CPM) is the endogenous pain relief mechanism responsible for the "pain-inhibits-pain" phenomenon. This mechanism can be activated experimentally, and its efficiency evaluated by experimental pain tests. According to the "pain-inhibits-pain" principle, during such an experimental testing paradigm, a painful test stimulus is typically applied, followed by a conditioning stimulus. The effect of the conditioning stimulus on the test stimulus is examined to determine whether or not the conditioning stimulus elicits an inhibitory effect. With this study, the investigators want to examine in pain-free adults whether and to what extend the efficacy of CPM is influenced by 1) attention (focus versus distraction), 2) intrinsic expectations (pain reduction versus no change versus pain increase) with regard to pain due to the CPM paradigm used, and 3) the order of application of the test stimulus and conditioning stimulus (sequential versus parallel paradigm).

DETAILED DESCRIPTION:
Despite the widespread use of CPM by researchers, there is still no gold standard for conducting this test. Both a sequential and a parallel application of the test stimulus and the conditioning stimulus are often used interchangeably and side by side. In both paradigms, the pain intensity or pain threshold of the test stimulus is first determined. Subsequently, in the parallel protocol, the test stimulus is reapplied while simultaneously applying the conditioning stimulus. In the sequential protocol, the conditioning stimulus is applied first, and after removing the latter stimulus, the test stimulus is reapplied (the CPM effect is visible up to 5 minutes after removal of the conditioning stimulus). The difference between the initial and repeated test stimulus (during or after conditioning) is quantified to express the CPM effect.

Even the publication of an expert opinion, which decided in favor of the sequential paradigm, has so far changed little in the use of the two paradigms. In that same publication, international CPM experts considered the sequential order 'purer' than the parallel order, as the results of the latter can be attributed to a shift of attention to the conditioning stimulus. However, this claim has little support from the literature. Some researchers even argue that cognitive mechanisms such as attentional shift might be part of the underlying mechanism of the CPM effect. Existing research also shows that CPM effectiveness is influenced by expectations. For this, previous studies conditioned test subjects by telling them in advance that the conditioning stimulus would reduce or increase pain. However, when the experimental CPM paradigm is used to investigate the effectiveness of the pain-inhibiting system, no such suggestions are made. However, this does not preclude that when the test protocol is explained to the subject, he or she does not create intrinsic expectations regarding the pain that is provoked. However, few studies have investigated this and the results of these studies are inconsistent and therefore do not allow conclusions to be drawn.

The aim of this study is to compare a sequential protocol with a parallel protocol on the one hand, and to measure the influence of expectations, attention and distraction on the CPM effect on the other.

In this study, the test stimulus of the CPM measurement will consist of a mechanical stimulus applied with an analog algometer (Force Dial model FDK 10 and 40 Push Pull Force Gage, Wagner instruments, Greenwich, Connecticut) on the Brachioradialis and Quadriceps muscle of the dominant side. The pressure pain threshold will be determined and used as an outcome measure. The conditioning stimulus consists of immersing the hand (up to 10 cm above the wrist) of the non-dominant side in warm water at a temperature of 45,5°C for 6 minutes. This temperature has been proven to be a reliable stimulus, eliciting solid effects.

At the time of testing, the CPM measurement will therefore be performed four times, each time with a small variation. The order of the variations is determined at random. There is a break of 10 minutes between each performance, so that the effect of the previous performance has worn off. The four variations of the CPM paradigm are the following:

1. Sequential protocol: the test stimulus is applied before and after the conditioning stimulus
2. Parallel protocol: the test stimulus is applied before, after and during immersion (at minute 4)
3. Focus protocol: this protocol works like the sequential protocol. In addition, the subject will be asked to give a pain score from 0 (no pain) to 100 (excruciating pain) every 30 seconds during immersion, thereby focusing on the conditioning stimulus.
4. Distraction protocol: this protocol works like the sequential protocol. During the immersion, attention will be diverted away from the conditioning stimulus by having the subject perform a cognitive test known as the Paced Auditory Serial Addition Test (PASAT). The latter implies that the subject must listen to an auditory series of numbers, memorize them and add them.

Before the actual test begins, a familiarization moment will take place, in which the subject becomes acquainted with the test and the conditioning stimulus by undergoing it for the first time. There will also be a practice session of the PASAT at that time.

Before the start of the CPM test, two questionnaires are taken: a general questionnaire assessing sociodemographic and health-related characteristics, and the Hospital Anxiety and Depression Scale (HADS), which provides an indication of feelings of anxiety and depression that the subject might experience, as such factors may have an influence (i.e. known confounders) on the CPM effect.

Finally, for each variation on the CPM paradigm, it will be briefly explained what the protocol to be undergone entails. This involves assessing the subject's expectations with regard to the related protocol. The subject will have to indicate whether he / she expects the immersion to have an influence on the pressure threshold measurement (yes, pain increase; yes, pain reduction; no, no effect). If the participants answer "yes", the subjects are asked to quantify the expected impact by indicating how much more or less pressure is expected to be tolerated (in percentages).

This study has a cross-sectional design and the familiarization and the experimental CPM assessments take place during during a single test session of about 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking participants (age between 18 and 65 years)
* Healthy volunteers who have no pain complaints

Exclusion Criteria:

* Not speaking Dutch
* A history of serious health issues (e.g. cancer, stroke, epilepsy, diabetes, depression, etc...)
* History of pain complaints or current pain (e.g. people who suffer from severe migraine, low back pain, neck pain, frozen shoulder, meniscectomy,...)
* Cognitive, arithmetic or attention disorders
* Pregnancy or breastfeeding in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy pain-free Dutch-speaking men and women between the age of 18 and 65 years. Participants will be recruited amongst friends, relatives and fellow students of the researchers.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) magnitude (kg/cm²) | cross-sectional (single test session, day 0)
  CPM magnitude is evaluated during 4 different CPM test protocols (sequential, focus, distraction, parallel) and will be compared between these protocols to answer the research questions. The test stimulus (i.e. mean mechanical pain pressure threshold measured at the Brachioradialis and Quadriceps muscle of the dominant side expressed in kg/cm²) is assessed before the application (minute 0) of the conditioning stimulus (i.e. hot thermal water immersion of the hand), and once again at minute 4 during conditioning stimulation (parallel protocol) or at 6 minutes 30 seconds which is 30 seconds after removal of the conditioning stimulus (sequential, focus and distraction protocol). CPM (kg/cm²) magnitude is calculated by subtracting the first test stimulus from the second test stimulus assessment, with a negative CPM value (kg/cm²) denoting pain inhibition, and a positive CPM (kg/cm²) value denoting pain facilitation.

SECONDARY OUTCOMES:
Sociodemographic and health-related characteristics | cross-sectional (single test session, day 0)
  A general questionnaire assessing sociodemographic and health related characteristics
Hospital Anxiety and Depression Scale (HADS) | cross-sectional (single test session, day 0)
  A questionnaire assessing anxiety and depression;
  A score on the subscale of: 0-7 (no anxiety disorder or depression), 8-10 (a possible anxiety disorder or depression), 11-21 (a suspected anxiety disorder or depression)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Prof, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Dept. of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] Goffaux P, Redmond WJ, Rainville P, Marchand S. Descending analgesia--when the spine echoes what the brain expects. Pain. 2007 Jul;130(1-2):137-43. doi: 10.1016/j.pain.2006.11.011. Epub 2007 Jan 9. PMID 17215080
- [Background] Bjorkedal E, Flaten MA. Expectations of increased and decreased pain explain the effect of conditioned pain modulation in females. J Pain Res. 2012;5:289-300. doi: 10.2147/JPR.S33559. Epub 2012 Aug 17. PMID 23049277
- [Background] Lewis GN, Leys A, Rice DA, McNair PJ. Subconscious manipulation of pain expectation can modulate cortical nociceptive processing. Pain Pract. 2015 Feb;15(2):117-23. doi: 10.1111/papr.12157. Epub 2013 Dec 11. PMID 24325269
- [Background] Cormier S, Piche M, Rainville P. Expectations modulate heterotopic noxious counter-stimulation analgesia. J Pain. 2013 Feb;14(2):114-25. doi: 10.1016/j.jpain.2012.10.006. Epub 2012 Dec 20. PMID 23260452
- [Background] France CR, Burns JW, Gupta RK, Buvanendran A, Chont M, Schuster E, Orlowska D, Bruehl S. Expectancy Effects on Conditioned Pain Modulation Are Not Influenced by Naloxone or Morphine. Ann Behav Med. 2016 Aug;50(4):497-505. doi: 10.1007/s12160-016-9775-y. PMID 26809850
- [Background] Kennedy DL, Kemp HI, Ridout D, Yarnitsky D, Rice ASC. Reliability of conditioned pain modulation: a systematic review. Pain. 2016 Nov;157(11):2410-2419. doi: 10.1097/j.pain.0000000000000689. PMID 27559835
- [Background] Nir RR, Granovsky Y, Yarnitsky D, Sprecher E, Granot M. A psychophysical study of endogenous analgesia: the role of the conditioning pain in the induction and magnitude of conditioned pain modulation. Eur J Pain. 2011 May;15(5):491-7. doi: 10.1016/j.ejpain.2010.10.001. Epub 2010 Oct 28. PMID 21035364
- [Background] Nir RR, Yarnitsky D, Honigman L, Granot M. Cognitive manipulation targeted at decreasing the conditioning pain perception reduces the efficacy of conditioned pain modulation. Pain. 2012 Jan;153(1):170-176. doi: 10.1016/j.pain.2011.10.010. Epub 2011 Nov 25. PMID 22119318
- [Background] Reinert A, Treede R, Bromm B. The pain inhibiting pain effect: an electrophysiological study in humans. Brain Res. 2000 Apr 17;862(1-2):103-10. doi: 10.1016/s0006-8993(00)02077-1. PMID 10799674
- [Background] Gronwall DM. Paced auditory serial-addition task: a measure of recovery from concussion. Percept Mot Skills. 1977 Apr;44(2):367-73. doi: 10.2466/pms.1977.44.2.367. PMID 866038
- [Background] Rao SM, Leo GJ, Haughton VM, St Aubin-Faubert P, Bernardin L. Correlation of magnetic resonance imaging with neuropsychological testing in multiple sclerosis. Neurology. 1989 Feb;39(2 Pt 1):161-6. doi: 10.1212/wnl.39.2.161. PMID 2915783
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Derived] Billens A, Dhondt E, Dierickx E, Van Damme S, De Greef I, Van Oosterwijck S, Meeus M, Van Oosterwijck J. Attentional Focus but Not Distraction or Expectations Influence Conditioned Pain Modulation in Healthy Adults. Eur J Pain. 2025 Jul;29(6):e70058. doi: 10.1002/ejp.70058. PMID 40542602